CLINICAL TRIAL: NCT00721123
Title: Long-term Extension Study of Safety During Treatment With Tocilizumab (MRA) in Patients Completing Treatment in WA17822
Brief Title: A Long-term Extension Study of Tocilizumab (Myeloma Receptor Antibody [MRA]) in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA18695
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab 8 mg/kg (Experimental): All participants received tocilizumab 8 mg/kg to a maximum of 800 mg, administered by intravenous (IV) infusion over one hour, every 4 weeks. Concomitant therapies were limited to dosage and administration constraints detailed in the protocol.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab (myeloma receptor antibody [MRA]) was supplied in sterile solution of 20 mg TCZ/mL for aseptic preparation of infusion bags for IV administration.
  Other Names: RoActemra; Actemra; Tocilizumab (MRA); TCZ

SUMMARY:
This open-label, international multi-center extension study WA18695 was designed to assess the long term safety of tocilizumab in patients who had moderate to severe active rheumatoid arthritis (RA). Patients enrolled in the WA18695 study had previously received treatment in the 24-week, placebo-controlled, Phase III Study WA17822. Eligible patients were assigned to treatment with 8 mg/kg tocilizumab every 4 weeks for a maximum of 5 years.

DETAILED DESCRIPTION:
The primary objective of this extension study was to assess the long-term safety of 8 mg/kg tocilizumab with regard to adverse events (AEs) and laboratory result abnormalities.

The secondary objectives were as follows:

* To explore the possibility of reducing concomitant steroid treatment
* To determine the long-term efficacy of 8 mg/kg tocilizumab with regard to reduction in signs and symptoms
* To better understand and predict tocilizumab efficacy, response, safety, and progression of rheumatoid arthritis (RA) and associated diseases with regard to its effect on biomarkers

No viable biomarkers for TCZ treatment effects were identified from the controlled studies. There were, therefore, no biomarkers that warranted further investigation in long-term studies, so no biomarker data are reported.

The extension study WA18695 was an open-label, international multi-center study in patients with moderate to severe active rheumatoid arthritis (RA) who had completed treatment in the 24 weeks placebo-controlled Phase III study WA17822. Patients entering WA17822 had an inadequate response to methotrexate (MTX), and, during WA17822, patients had received treatment with intravenous infusions of tocilizumab 4 mg/kg, 8 mg/kg, or placebo every 4 weeks with background MTX therapy.

All patients who completed the planned course of treatment or escape therapy in the WA17822 study were eligible to enter the WA18695 long-term extension study, where they were assigned to treatment with 8 mg/kg RoActemra/Actemra plus MTX. The dose of RA medications such as MTX and nonsteroidal anti-inflammatory drugs (NSAIDs), but excluding corticosteroids, was to be kept stable for the first 48 weeks of the WA18695 study. During this time dose reductions in these treatments were only allowed as clinically required for safety reasons. After week 48, the administration of disease-modifying antirheumatic drugs (DMARDs) and NSAIDs could be changed, according to the investigator's practice and as tolerated by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed participation in the Phase III study WA17822 (NCT00106548) in adult rheumatoid arthritis.

Exclusion Criteria:

* Treatment with any investigational agent since the last administration of study drug in WA17822.
* Treatment with intravenous (IV) gammaglobulin, plasmapheresis, or Prosorba column since the last administration of study drug in WA17822.
* Treatment with an anti-tumor necrosis factor or anti-interleukin-1 agent, or a T cell costimulation modulator since the last administration of study drug in WA17822.
* Previous treatment with any cell-depleting therapies.
* Parenteral, intramuscular, or intra-articular corticosteroids within 6 weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2005-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- Buenos Aires, Argentina
- Australia (3):
  - Adelaide
  - Maroochydore
  - Shenton Park
- Vienna, Austria
- Brazil (2):
  - Porto Alegre
  - São Paulo
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (10):
  - Calgary, Alberta
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- France (4):
  - Besançon
  - Créteil
  - Le Mans
  - Paris
- Germany (7):
  - Bad Bramstedt
  - Bad Nauheim
  - Baden-Baden
  - Berlin
  - Cologne
  - Erlangen
  - Heidelberg
- Hong Kong (2):
  - Hong Kong
  - Tuenmen
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (5):
  - Cona (ferrara)
  - Gazzi
  - Palermo
  - Siena
  - Udine
- Mexico (5):
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - México
  - San Luis Potosí City
- Singapore, Singapore
- Piešťany, Slovakia
- Switzerland (2):
  - Bern
  - Lausanne
- Thailand (2):
  - Bangkok
  - Chiang Mai

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 mg/kg: Patients received tocilizumab (TCZ) 8 mg/kg intravenously every 4 weeks.
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg
Started | 538
Completed | 355
Not Completed | 183
Not completed — Adverse Event | 96
Not completed — Death | 10
Not completed — Insufficient Therapeutic Response | 21
Not completed — Protocol Violation | 1
Not completed — Refused Treatment | 41
Not completed — Failure to Return | 9
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All-exposure population: All patients who entered the study and received at least one dose of tocilizumab at any time. Baseline was defined as the first dose of study drug, whether that occurred in the WA17822 study or the WA18695 study.
Groups:
- Tocilizumab 8 mg/kg: Patients received tocilizumab 8 mg/kg intravenously every 4 weeks.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 538
Age Continuous [Mean (Standard Deviation); unit: years] | 50.8 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 443
  Male | 95

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event (AE) Summary Over Time
Description: The number of participants experiencing at least one adverse event (AE) is recorded for each 12-month time period, with multiple occurrences in a single individual counted. Because months were calculated as 28 days, the periods actually equate to 48 weeks.
Time Frame: through 264 Weeks
Population: All exposure population, which includes all participants who entered the study and received at least one dose of tocilizumab at any time.
Measure: Number; unit: Participants
Groups:
- Months 0 - 12: Participants with scores during Months 0-12, which equates to baseline through Week 48.
- Months 13 - 24: Participants with scores during Months 13 - 24, which equates to Weeks 49-96.
- Months 25 - 36: Participants with scores during Months 25 - 36, which equates to Weeks 97-144.
- Months 37 - 48: Participants with scores during Months 37 - 48, which equates to Weeks 145-192.
- Months Greater Than 48: Participants with scores during Months greater than 48, which equates to Weeks 193-264.
Arm/Group | Months 0 - 12 | Months 13 - 24 | Months 25 - 36 | Months 37 - 48 | Months Greater Than 48
Number analyzed (Participants) | 538 | 509 | 463 | 434 | 414
Participants
  Experienced an adverse event | 433 | 390 | 333 | 294 | 329
  Experienced a serious adverse event | 55 | 55 | 55 | 35 | 74
  Experienced AE leading to withdrawal | 24 | 17 | 22 | 8 | 32

2. Secondary Outcome: Participants Showing Improvement in Rheumatoid Arthritis Symptoms Over Time, Through 264 Weeks
Description: The American College of Rheumatology (ACR) established certain criteria to measure improvement in rheumatoid arthritis symptoms that include tender or swollen joint counts and five other criteria, including acute phase reactant, patient assessment, physician assessment, pain scale, and disability/functional questionnaire.
  Clinical trials use the ACR Score, based on those criteria, as a standard for reporting different degrees of improvement in rheumatoid arthritis symptoms.
  Scores on the ACR scale may be up to ACR100 because the number after "ACR" is the percent of improvement in tender or swollen joint counts as well as in three of the other five criteria. Clinical trials determine the percentage of participants who achieve that score - that percentage of improvement.
Time Frame: through 264 Weeks
Population: All exposure population, which includes all participants who entered the study and received at least one dose of tocilizumab, with a score at the given time point.
Measure: Number; unit: Percentage of Participants
Groups:
- Week 24: Participants with scores at 24 weeks post-baseline.
- Week 48: Participants with scores at 48 weeks post-baseline.
- Week 108: Participants with scores at 108 weeks post-baseline.
- Week 156: Participants with scores at 156 weeks post-baseline.
- Week 204: Participants with scores at 204 weeks post-baseline.
- Week 264: Participants with scores at 264 weeks post-baseline.
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 522 | 480 | 422 | 413 | 387 | 367
Percentage of Participants
  ACR20 | 63.2 | 76.0 | 81.2 | 83.3 | 82.2 | 83.9
  ACR50 | 41.2 | 50.6 | 58.1 | 59.6 | 62.5 | 67.8
  ACR70 | 17.4 | 27.1 | 38.2 | 41.9 | 42.1 | 45.8
  ACR90 | 4.8 | 5.2 | 11.3 | 15.3 | 16.8 | 19.3

3. Secondary Outcome: Percentage of Participants Classified as Responders by Disease Activity Scores Over Time, Through 264 Weeks
Description: The disease activity score 28 (DAS28) is a combined index for measuring disease activity in rheumatic arthritis (RA) that includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The DAS28 scale ranges from 0 to 10, where lower scores represent less disease activity. Participants with DAS28 scores less than 2.6 were categorized as responders with remission and those with DAS 28 scores of 3.2 or less were categorized as responders with low disease activity (LDA). The percentage of participants classified as responders in each category was recorded over time.
Time Frame: through 264 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 516 | 470 | 430 | 410 | 381 | 363
Percentage of Participants
  Responders with Remission (DAS<2.6) | 24.6 | 43.0 | 53.7 | 54.9 | 57.2 | 60.6
  Responders with Low Disease Activity (DAS</= 3.2) | 41.7 | 57.7 | 67.0 | 71.2 | 70.6 | 72.2

4. Secondary Outcome: Percentage of Participants Classified as Responders by EULAR Response Over Time, Through 264 Weeks
Description: Participants were classified as responders based on a European League Against Rheumatism (EULAR) response of Good or Moderate. Comparing the DAS28 from one patient on two different time points, it is possible to define improvement or response. The EULAR response criteria take into consideration both the first score and the change in score in order to classify them as good response, moderate response or no response. The percentage of participants who were classified as responders was recorded, as posted below.
Time Frame: through 264 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 514 | 468 | 429 | 409 | 380 | 362
Percentage of Participants
  EULAR Good Response | 41.2 | 56.6 | 65.5 | 70.9 | 69.5 | 71.0
  EULAR Moderate Response | 48.1 | 39.1 | 29.8 | 25.9 | 26.8 | 25.1

5. Secondary Outcome: Change From Baseline in Scores for Swollen and Tender Joint Counts Over Time, Through 264 Weeks
Description: Swollen joint count (SJC) includes an assessment of 66 joints, and tender joint count (TJC) include an assessment of 68 joints. Joint prosthesis, arthrodesis or fused joints were not considered. Joints were assessed and classified as swollen/not swollen, and tender/not tender, by pressure and joint manipulation on physical examination. Change from Baseline in the SJC and TJC were calculated at given time points, and a negative change indicates improvement.
  A small proportion of participants in the all-exposure population reduced or stopped their oral corticosteroid use due to sustained efficacy (defined as at least a 50% improvement in both swollen joint count (SJC) and tender joint count (TJC).
Time Frame: through 264 Weeks
Population: All exposure population, which includes all participants who entered the study and received at least one dose of tocilizumab at any time, with a score at the given time point.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 532 | 506 | 454 | 422 | 405 | 371
Joints
  Swollen Joint Count (SJC) | -11.7 (11.50) | -13.6 (11.04) | -15.6 (11.51) | -16.2 (11.46) | -16.2 (11.48) | -16.5 (11.26)
  Tender Joint Count (TJC) | -17.4 (14.82) | -20.3 (15.12) | -23.1 (15.82) | -23.8 (16.14) | -23.8 (15.89) | -24.8 (16.37)

6. Secondary Outcome: Change From Baseline in Scores for Health Assessment Questionnaire - Disability Index Over Time, Through 264 Weeks
Description: The Stanford Health Assessment Questionnaire - Disability Index (HAQ-DI) is a questionnaire specific for rheumatoid arthritis with 8 component sets (domains): dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each domain has 2-3 questions (for a total of 20) that participants answer with categorical answers enumerated as a scale of 0-3, where 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do.
  To calculate the HAQ-DI the patient must have a domain score for at least 6 of the eight domains. The HAQ-DI is the sum of the domain scores, divided by the number of domains that have a score (in range 6-8). The resulting HAQ-DI scores are on a scale that ranges from 0 to 3, where 0=lowest level of difficulty and 3=highest level of difficulty. A negative change from baseline indicates improvement.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 445 | 408 | 376 | 349 | 332 | 316
Units on a Scale | -0.49 (0.582) | -0.53 (0.614) | -0.59 (0.636) | -0.61 (0.655) | -0.65 (0.661) | -0.62 (0.693)

7. Secondary Outcome: Change From Baseline in Scores for Patient's Global Assessment of Disease Activity Over Time, Through 264 Weeks
Description: Patient's global assessment of disease activity is the patient's overall assessment of their disease activity during specified time periods on a 100 mm horizontal visual analogue scale (VAS). The left-hand extreme of the line was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme as "maximum disease activity" (maximum arthritis disease activity). Change from baseline was calculated for given periods, and a negative change indicates improvement.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 521 | 479 | 442 | 414 | 387 | 367
Units on a Scale | -26.6 (26.87) | -30.3 (27.71) | -31.1 (27.65) | -31.6 (26.74) | -33.0 (26.83) | -32.9 (27.58)

8. Secondary Outcome: Change From Baseline in Scores for Physician's Global Assessment of Disease Activity Over Time, Through 264 Weeks
Description: Physician's global assessment of disease activity is the treating physician's assessment of the patient's current disease activity on a 100 mm horizontal visual analogue scale (VAS). The extreme left end of the line was described as "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end as "maximum disease activity". Change from baseline was calculated for given periods, and a negative change indicates improvement.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 521 | 479 | 439 | 416 | 389 | 369
Units on a Scale | -33.8 (23.33) | -38.1 (23.77) | -41.1 (23.79) | -43.2 (23.26) | -44.8 (22.66) | -44.4 (23.64)

9. Secondary Outcome: Change From Baseline in Scores for Patient's Level of Pain Over Time, Through 264 Weeks
Description: The patient's assessment of the patient's current level of pain on a 100 mm horizontal VAS was recorded. The extreme left end of the line was described as "no pain" and the extreme right end as "unbearable pain". Change from baseline was calculated for given periods, and a negative change indicates improvement.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 521 | 479 | 442 | 414 | 388 | 367
Units on a Scale | -23.7 (26.38) | -26.7 (27.27) | -28.0 (26.33) | -28.1 (25.99) | -29.5 (26.98) | -29.2 (26.84)

10. Primary Outcome: Summary Adverse Event Rates Over Time
Description: Patient year (PY) refers to duration in study, calculated from first active drug intake to last safety assessment available + 1. Patient year rates with confidence interval were calculated for adverse events of interest in evaluating the long-term safety of the product being studied.
  Abbreviations include the following: adverse event (AE), adverse event of special interest (AESI), gastrointestinal (GI), serious adverse event (SAE), and investigational product (IP). Hypersensitivity events were defined as AEs that occurred during or within 24 hours of IP infusion and were not deemed "unrelated" to trial treatment by the investigator. This definition includes all types of AEs, regardless of whether or not they were consistent with hypersensitivity.
  Medical confirmation of the AESI "GI perforation" was based on medical adjudication of events captured by the GI Perforation Standardised MedDRA Queries (SMQs).
Time Frame: through 264 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Adverse Events per 100 Patient Years
Groups:
- Months 0 - 12: Participants with scores during Months 0-12, which equates to baseline through Week 48 (Total PY=486.34).
- Months 13 - 24: Participants with scores during Months 13 - 24, which equates to Weeks 49-96 (Total PY=444.49).
- Months 25 - 36: Participants with scores during Months 25 - 36, which equates to Weeks 97-144 (Total PY=410.93).
- Months 37 - 48: Participants with scores during Months 37 - 48, which equates to Weeks 145-192 (Total PY=388.25).
- Months Greater Than 48: Participants with scores during Months greater than 48, which equates to Weeks 193-264 (Total PY=731.93).
Arm/Group | Months 0 - 12 | Months 13 - 24 | Months 25 - 36 | Months 37 - 48 | Months Greater Than 48
Number analyzed (Participants) | 538 | 509 | 463 | 434 | 414
Adverse Events per 100 Patient Years
  Total AE rate | 393.76 [376.32 to 411.80] | 286.17 [270.66 to 302.34] | 260.14 [244.78 to 276.22] | 249.84 [234.36 to 266.07] | 212.04 [201.62 to 222.86]
  Total SAE rate | 12.54 [9.59 to 16.11] | 13.05 [9.91 to 16.87] | 18.74 [14.79 to 23.42] | 12.62 [9.34 to 16.69] | 13.12 [10.62 to 16.02]
  Rate for AEs leading to withdrawal | 5.14 [3.33 to 7.59] | 3.82 [2.23 to 6.12] | 5.35 [3.36 to 8.11] | 2.06 [0.89 to 4.06] | 4.37 [2.99 to 6.17]
  AESI All Infections | 92.94 [84.57 to 101.92] | 87.52 [79.03 to 96.66] | 87.36 [78.56 to 96.88] | 87.32 [78.27 to 97.12] | 72.82 [66.77 to 79.27]
  AESI Serious Infections | 3.29 [1.88 to 5.34] | 2.47 [1.24 to 4.43] | 5.60 [3.55 to 8.40] | 3.35 [1.78 to 5.73] | 3.55 [2.32 to 5.20]
  AESI Opportunistic infections | 0 [NA to NA] — There were no opportunistic infections in this period. | 0.22 [0.01 to 1.25] | 0 [NA to NA] — There were no opportunistic infections in this period. | 0.52 [0.06 to 1.86] | 0.27 [0.03 to 0.99]
  AESI Hypersensitivity events | 27.35 [22.90 to 32.41] | 9.90 [7.19 to 13.29] | 5.35 [3.36 to 8.11] | 3.86 [2.16 to 6.37] | 4.10 [2.77 to 5.85]
  AESI Hepatic events | 0.41 [0.05 to 1.49] | 0.90 [0.25 to 2.30] | 0.49 [0.06 to 1.76] | 1.03 [0.28 to 2.64] | 0.68 [0.22 to 1.59]
  AESI Myocardial infarction | 0.62 [0.13 to 1.80] | 0 [NA to NA] — There were no myocardial infarctions in this period. | 0.24 [0.01 to 1.36] | 0.77 [0.16 to 2.26] | 0.27 [0.03 to 0.99]
  AESI Stroke, ischemic or hemorrhagic | 0.21 [0.01 to 1.15] | 0.22 [0.01 to 1.25] | 0.73 [0.15 to 2.13] | 0.26 [0.01 to 1.44] | 0.41 [0.08 to 1.20]
  AESI GI perforation | 0 [NA to NA] — There were no medically confirmed GI perforations in this period. | 0 [NA to NA] — There were no medically confirmed GI perforations in this period. | 0.49 [0.06 to 1.76] | 0.26 [0.01 to 1.44] | 0 [NA to NA] — There were no medically confirmed GI perforations in this period.
  AESI Malignancy | 1.23 [0.45 to 2.69] | 1.80 [0.78 to 3.55] | 0.97 [0.27 to 2.49] | 0.77 [0.16 to 2.26] | 1.50 [0.75 to 2.69]
  AESI Demyelinating disorders | 0.21 [0.01 to 1.15] | 0 [NA to NA] — There were no demyelinating disorders in this period. | 0 [NA to NA] — There were no demyelinating disorders in this period. | 0 [NA to NA] — There were no demyelinating disorders in this period. | 0 [NA to NA] — There were no demyelinating disorders in this period.
  AESI Serious bleeding disorders | 0.62 [0.13 to 1.80] | 0.45 [0.05 to 1.63] | 0.49 [0.06 to 1.76] | 0.26 [0.01 to 1.44] | 0.68 [0.22 to 1.59]

11. Primary Outcome: Overall Death Rate Over Time
Description: Patient year (PY) refers to duration in study, calculated from first active drug intake to last safety assessment available + 1.
  To calculate the death rate, the total cumulative number of years that all participants were exposed to the drug, from first active drug intake to last safety assessment available + 1, was calculated as 2461.94. Since 10 participants died during that time, the death rate per year was not informative (0.00). Therefore, the overall death rate was calculated with the confidence interval based on events per 100 patient years exposure.
Time Frame: through 264 Weeks
Population: All exposure population, which included all participants who entered the study and received at least one dose of tocilizumab at any time.
Measure: Number (95% Confidence Interval); unit: Deaths per 100 PY
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 538
Deaths per 100 PY | 0.41 [0.19 to 0.75]

12. Secondary Outcome: Percentage of Participants With at Least a 5-point Improvement From Baseline in Quality of Life Measure for Fatigue Over Time, Through 264 Weeks
Description: Quality of life is measured using the sub-scale for Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). The assessment was originally developed for chronic illnesses and is now widely used for patients with rheumatoid arthritis.
  FACIT-F is a 13-item questionnaire. Participants score each item on a 5-point scale: 0 (Not at all) to 4 (Very much), for a highest possible score of 52. The responses are transformed into a FACIT-F score, where a higher score reflects an improvement. The percentage of participants with at least a 5-point improvement from baseline in the Facit-F score is shown at categorical time points.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 523 | 482 | 444 | 414 | 390 | 370
Percentage of Participants | 66.0 | 58.7 | 61.5 | 62.3 | 60.0 | 62.2

13. Secondary Outcome: Percentage of Participants With at Least a 5-point Improvement From Baseline in Quality of Life Using the 36-Item Short-Form Health Survey (SF-36) Over Time, Through 264 Weeks
Description: The SF-36 Health Survey is a standardized questionnaire consisting of 36 questions that measures patient-reported symptoms on 8 dimensions; it is used to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100. A positive change score indicates better HRQoL. The percentage of participants with at least a 5-point improvement from baseline is presented for each subscale.
Time Frame: through 264 Weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Week 24 | Week 48 | Week 108 | Week 156 | Week 204 | Week 264
Number analyzed (Participants) | 423 | 424 | 395 | 373 | 344 | 334
Percentage of Participants
  SF-36 MCS | 48.2 | 46.2 | 48.6 | 49.9 | 49.7 | 49.1
  SF-36 PCS | 63.8 | 69.1 | 71.1 | 71.3 | 73.3 | 71.3

ADVERSE EVENTS:
Description: All-exposure population: All patients who entered the study and received at least 1 dose of tocilizumab at any time.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 199/538
Other Adverse Events (participants affected / at risk) | 475/538
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=538)
Pneumonia (Infections and infestations) | 12
Diverticulitis (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 4
Erysipelas (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 4
Abscess limb (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Cellulitis staphylococcal (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Pneumonia pneumococcal (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 2
Varicella (Infections and infestations) | 2
Abscess neck (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bursitis infective staphylococcal (Infections and infestations) | 1
Douglas' abscess (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung Abscess (Infections and infestations) | 1
Mediastinitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Proteus infection (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Septic arthritis (Infections and infestations) | 1
Staphylococcal septic shock (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer state unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Fractured ischium (Injury, poisoning and procedural complications) | 1
Gas poisoning (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Inguinal hernia (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Diverticular perforation (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Dressler's syndrome (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Sciatica (Nervous system disorders) | 3
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Essential tremor (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 3
Vericose vein (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Iliac artery occlusion (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Vasculitis necrotising (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 4
Cholelithiasis (Hepatobiliary disorders) | 4
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1
Perforation bile duct (Hepatobiliary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1
Confusional state (Psychiatric disorders) | 2
Adjustment disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 2
Uterine haemorrhage (Reproductive system and breast disorders) | 2
Endometriosis (Reproductive system and breast disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Device breakage (General disorders) | 2
Device dislocation (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Chest pain (General disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3
Cataract (Eye disorders) | 2
Ulcerative keratitis (Eye disorders) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=538)
Upper respiratory tract infection (Infections and infestations) | 136
Nasopharyngitis (Infections and infestations) | 133
Urinary tract infection (Infections and infestations) | 93
Bronchitis (Infections and infestations) | 83
Gastroenteritis (Infections and infestations) | 69
Pharyngitis (Infections and infestations) | 60
Influenza (Infections and infestations) | 43
Oral herpes (Infections and infestations) | 37
Sinusitis (Infections and infestations) | 32
Rhinitis (Infections and infestations) | 31
Diarrhoea (Gastrointestinal disorders) | 85
Dyspepsia (Gastrointestinal disorders) | 85
Nausea (Gastrointestinal disorders) | 50
Gastritis (Gastrointestinal disorders) | 35
Abdominal pain (Gastrointestinal disorders) | 32
Abdominal pain upper (Gastrointestinal disorders) | 32
Mouth ulceration (Gastrointestinal disorders) | 29
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 28
Back pain (Musculoskeletal and connective tissue disorders) | 64
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 64
Arthralgia (Musculoskeletal and connective tissue disorders) | 37
Headache (Nervous system disorders) | 89
Dizziness (Nervous system disorders) | 35
Hypertension (Vascular disorders) | 107
Alanine aminotransferase increased (Investigations) | 59
Transaminases increased (Investigations) | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 46
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32
Depression (Psychiatric disorders) | 43
Insomnia (Psychiatric disorders) | 30
Hypercholesterolaemia (Metabolism and nutrition disorders) | 33
Leukopenia (Blood and lymphatic system disorders) | 31
Rash (Skin and subcutaneous tissue disorders) | 30
Vertigo (Ear and labyrinth disorders) | 27
Conjunctivitis (Eye disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.